CLINICAL TRIAL: NCT03789695
Title: RE-ELECT Study: "Randomized Evaluation of Changing Kidney Function Over a Time in Patients With Atrial Fibrillation (AF), Concomitant T2DM and Existing Chronic Kidney Disease (CKD) Treated With Dabigatran or Warfarin for Stroke Prevention"
Brief Title: RE-ELECT. Dabigatran vs Warfarin in AF Patients With T2DM and CKD
Acronym: RE-ELECT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Irina Ermolaeva (Other)
Responsible Party: Sponsor-Investigator, Irina Ermolaeva, Head of Department of preclinical and clinical trials management, I.M. Sechenov First Moscow State Medical University
Organization: I.M. Sechenov First Moscow State Medical University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1160.283
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation; T2DM (Type 2 Diabetes Mellitus); Chronic Kidney Diseases
MeSH Terms: conditions — Atrial Fibrillation; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Dabigatran

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dabigatran etexilate (Experimental): Dabigatran etexilate (Pradaxa) 110 mg b.i.d. or 150 mg b.i.d. according SmPC during 2 years
  Interventions: Drug: Dabigatran Etexilate
- Warfarin (Active Comparator): Warfarin under the control of INR once a month (target range 2.0 - 3.0) during 2 years
  Interventions: Drug: Dabigatran Etexilate

INTERVENTIONS:
Drug: Dabigatran Etexilate — Study drug dabigatran etexilate. There are two dosage regimens of dabigatran etexilate used in the study: 150 mg b.i.d. and 110 mg b.i.d. The dose of dabigatran etexilate will be chosen by the investigator in accordance with Russian PRADAXA SmPC
  Other Names: Pradaxa

SUMMARY:
Kidney function in patients with atrial fibrillation (AF) is tending to decline over a time which is clearly demonstrated in clinical studies. Renal impairment is a risk factor for stroke, its progression is associated with unfavorable prognosis. So preserving kidney function should be considered as a one of priorities when choosing treatment strategies which is especially important in patients with existing chronic kidney disease (CKD) or in patients who have risk of its development. This is especially relevant for the patients with type 2 diabetes mellitus (T2DM) and with CKD who can be considered as a group of risk for rapid kidney function decline.

DETAILED DESCRIPTION:
It is suggested that the decline in renal function may occur more slowly in patients receiving dabigatran etexilate (Pradaxa) compared to patients taking warfarin. The planned trial is a prospective phase IV randomized trial in which patients with AF, T2DM and CKD will be randomized to groups receiving either dabigatran etexilate (Pradaxa) or warfarin. The main goal of the study is to assess the differences in annual eGFR reduction between patients receiving dabigatran etexilate (Pradaxa) or warfarin for 24 months. The difference in annual eGFR reduction will be estimated using the SMPI parameters (mixed model of repeated measurements). Secondary goals are as follows: - to evaluate the progression of albuminuria during treatment with dabigatran etexilate (Pradaxa) or warfarin based on the combined endpoint; - to evaluate the dynamics of the albumin/creatinine ratio (ACR) in urine during 2 years of treatment with dabigatran etexilate (Pradaxa) or warfarin; - to evaluate bleeding episodes, acute cerebrovascular accident, and systemic embolism in the dabigatran etexilate (Pradaxa) and warfarin groups; - to compare glycemic control (HbA1c) in patients receiving dabigatran etexilate (Pradaxa) and warfarin

ELIGIBILITY:
Inclusion Criteria:

* Non-valvular atrial fibrillation
* Diagnosis of T2D according to Russian Clinical Guidelines
* Chronic kidney disease according to KDIGO definition*
* Stable RAS background treatment
* Age > 18 yrs;
* Informed consent to participate in the study signed by the patient.

Exclusion Criteria:

* HbA1c >10%
* UACR > 3000
* Renal transplant
* Biopsy proven kidney entities other than Diabetic Kidney Disease (if known only, no kidney biopsy is planned within the study)
* Background immunosuppressant therapy
* Hematologic disorders which can influence hemostasis (hemoblastosis, etc.); connective tissue diseases (SLE, systemic scleroderma, dermatomyositis) and any vasculitis;
* Primary or secondary antiphospholipid syndrome;
* Known cancer diagnosis;
* Major surgical interventions within 3 months before the study enrollment and planned for the timelines of the study;
* Clinically relevant bleeding events within 3 months before the study enrollment;
* Acute coronary syndrome, PCI or CABG within 12 months before the study enrollment;
* Hemorrhagic stroke within 12 months before the study enrollment;
* Organ damages resulted from clinically relevant bleeding within 6 months before randomization
* Major trauma or any craniocerebral trauma within 30 days before randomization
* Uncontrolled hypertension (systolic BP>180 and or diastolic BP>100 while on antihypertensive treatment)
* CHF III-IV functional class (by NYHA)
* Ischemic stroke within the last 14 days before randomization
* Concomitant aspirin and/or clopidogrel use;
* Persistent use of drugs with potential nephrotoxic effects (NSAIDs, cytotoxic drugs etc.);
* Need in anticoagulation treatment for disease other than AF
* Pregnancy and lactation;
* Creatinine clearance < 30 ml/min (by Cockroft - Gault equation)
* Thrombocytopenia of <100 *109 /л
* Hepatic failure B and C by Child-Pugh score
* Psychiatrist disorders
* Background poor compliance
* Known hypersensitivity to dabigatran, warfarin or their components
* Life expectancy less than two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Difference in annual eGFR decline (slopes) between dabigatran and warfarin patients | 2 years
  * eGFR is to be calculated with CKD-EPI equation at baseline and at subsequent major visits.
  * for primary analysis only eGFR levels at one year and second year of treatment will be used. In case of one of values required for the analysis is missed LOCF (last observational carried forward) approach will be used

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Napalkov, Principal Investigator — First Moscow State Medical University (Sechenov's University)
Locations (1):
- I.M.Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No